CLINICAL TRIAL: NCT01156727
Title: Linking National Guard Veterans With Need to Mental Health Care
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDP 10-047
Record Dates: First submitted 2010-06-22; First posted 2010-07-05 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: OEF/OIF; Mental Health; Veterans
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- SURVEY: 6 months post-deployment: Michigan Army National Guard soldiers 6 months post deployment between August 2011 and December 2013
- SURVEY: 12 months post-deployment: Michigan Army National Guard soldiers 12 months post deployment between August 2011 and December 2013.
- INTERVIEWS: Michigan Army National Guard soldiers 12-24 months post deployment between October 2011-April 2014. Also key stakeholders from the B2B program.

SUMMARY:
This project added an evaluation/research component to an existing peer outreach program, implemented for over 1100 soldiers in the Michigan Army National Guard. The study aims were to: 1) evaluate the implementation of the B2B program to inform ongoing program modifications and facilitate future dissemination efforts, 2) assess whether the B2B program increases mental health and substance use treatment initiation and treatment retention among returning National Guard soldiers, and 3) explore whether the B2B program improves mental health symptoms, deceases hazardous alcohol use, and improves soldier well-being.

DETAILED DESCRIPTION:
The study aims were to: 1) evaluate the implementation of the B2B program to inform ongoing program modifications and facilitate future dissemination efforts, 2) assess whether the B2B program increases mental health and substance use treatment initiation and treatment retention among returning National Guard soldiers, and 3) explore whether the B2B program improves mental health symptoms, deceases hazardous alcohol use, and improves soldier well-being.

The study had three components which addressed each of the three specific aims. The first component assessed B2B implementation using an embedded mixed methods design. This evaluation included real-time assessment and adaptation of the program, as well as retrospective evaluation of implementation process, sustainability, and potential for spread. The second component addressed the impact of B2B on treatment initiation and retention. Preliminary analyses were completed using regression analyses. Pending additional data from the DoD, an interrupted time series design to assess Michigan National Guard soldiers' VA and non-VA services use in multiple time periods before and after the date of B2B implementation will be conducted.. The third study component assessed the impact of B2B on MI ARNG soldiers' outcomes using longitudinal survey data and adjusting for baseline mental health status using data from the Post Deployment Health Assessment (PDHA).

ELIGIBILITY:
Inclusion Criteria:

Michigan Army National Guard soldiers who have returned from OEF/OIF deployments between August 2010 and December 2012.

Exclusion Criteria:

Soldiers who did not return from deployment during the study time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SURVEY: Michigan Army National Guard soldiers who have returned from OEF/OIF deployments between August 2010 and December 2012.
  INTERVIEW: Michigan Army National Guard soldiers and key B2B stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 3015 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
Hazardous alcohol use | 6 and 12 months post deployment
  Hazardous alcohol use was assessed using the AUDIT-C, a 3-item alcohol screen for hazardous drinking and active alcohol use disorders (including alcohol abuse or dependence). In men, a score of 4 or more is considered positive, and in women, a score of 3 or more is considered positive.
PTSD symptoms | 6 and 12 months post deployment
  The PCL is a 17-item self-report checklist of PTSD symptoms based closely on the DSM-IV criteria. The PCL-M is a military version and questions refer to "a stressful military experience". Total possible scores range from 17 to 85. Higher scores indicate more symptoms of PTSD and a cut-off score of 50 is used for indicating a probable diagnosis of combat-related PTSD.
Depressive symptoms | 6 and 12 months post deployment
  The 21-item Beck Depression Inventory-2nd Edition (BDI-II) was used to assess depressive symptoms. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Awareness of B2B Program | 6 and 12 months post deployment
  National Guard soldiers were considered to be aware of the B2B program if they endorsed a survey item asking about awareness of the B2B program in the MIARNG. The question was, "I am aware that the MI ARNG has a B2B program," with response items of "No" and "Yes."

SECONDARY OUTCOMES:
Mental Health service utilization | 6 and 12 months post deployment
  National Guard soldiers were considered to have received mental health services if they endorsed any of 14 survey items asking about the receipt of mental health services for a stress, emotional, alcohol, or family problem from either general medical or mental health providers in a variety of settings (military, civilian, VA clinics, or in vet centers) in the last year. The question format used was "In the past, have you received mental health services for a stress, emotional, or family problem from: [specified provider] with response items of "No," "Yes, in the last year," or "Yes, but more than a year ago."

CONTACTS AND LOCATIONS:
Overall Officials: Marcia T. Valenstein, MD AB, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Valenstein M, Gorman L, Blow AJ, Ganoczy D, Walters H, Kees M, Pfeiffer PN, Kim HM, Lagrou R, Wadsworth SM, Rauch SA, Dalack GW. Reported barriers to mental health care in three samples of U.S. Army National Guard soldiers at three time points. J Trauma Stress. 2014 Aug;27(4):406-14. doi: 10.1002/jts.21942. PMID 25158634
- [Result] Bonar EE, Bohnert KM, Walters HM, Ganoczy D, Valenstein M. Student and Nonstudent National Guard Service Members/Veterans and Their Use of Services for Mental Health Symptoms. J Am Coll Health. 2015;63(7):437-46. doi: 10.1080/07448481.2014.975718. PMID 25337770
- [Result] Sripada RK, Richards SK, Rauch SA, Walters HM, Ganoczy D, Bohnert KM, Gorman LA, Kees M, Blow AJ, Valenstein M. Socioeconomic Status and Mental Health Service Use Among National Guard Soldiers. Psychiatr Serv. 2015 Sep;66(9):992-5. doi: 10.1176/appi.ps.201400346. Epub 2015 May 1. PMID 25930042
- [Result] Sripada RK, Bohnert AS, Teo AR, Levine DS, Pfeiffer PN, Bowersox NW, Mizruchi MS, Chermack ST, Ganoczy D, Walters H, Valenstein M. Social networks, mental health problems, and mental health service utilization in OEF/OIF National Guard veterans. Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1367-78. doi: 10.1007/s00127-015-1078-2. Epub 2015 Jun 2. PMID 26032182
- [Result] Nelson CB, Zivin K, Walters H, Ganoczy D, MacDermid Wadsworth S, Valenstein M. Factors Associated With Civilian Employment, Work Satisfaction, and Performance Among National Guard Members. Psychiatr Serv. 2015 Dec 1;66(12):1318-25. doi: 10.1176/appi.ps.201400334. Epub 2015 Aug 17. PMID 26278223
- [Result] Gorman LA, Sripada RK, Ganoczy D, Walters HM, Bohnert KM, Dalack GW, Valenstein M. Determinants of National Guard Mental Health Service Utilization in VA versus Non-VA Settings. Health Serv Res. 2016 Oct;51(5):1814-37. doi: 10.1111/1475-6773.12446. Epub 2016 Feb 3. PMID 26840993
- [Result] Zivin K, Yosef M, Levine DS, Abraham KM, Miller EM, Henry J, Nelson CB, Pfeiffer PN, Sripada RK, Harrod M, Valenstein M. Employment status, employment functioning, and barriers to employment among VA primary care patients. J Affect Disord. 2016 Mar 15;193:194-202. doi: 10.1016/j.jad.2015.12.054. Epub 2015 Dec 30. PMID 26773911
- [Result] Kim HM, Levine DS, Pfeiffer PN, Blow AJ, Marchiondo C, Walters H, Valenstein M. Postdeployment Suicide Risk Increases Over a 6-month Period: Predictors of Increased Risk among Midwestern Army National Guard Soldiers. Suicide Life Threat Behav. 2017 Aug;47(4):421-435. doi: 10.1111/sltb.12303. Epub 2016 Oct 5. PMID 27704587